CLINICAL TRIAL: NCT04886089
Title: Pre-anesthesia Pleth Variability Index as a Predictor for Post-induction Hypotension in Elderly Patients Undergoing General Anesthesia: A Prospective Cohort Study
Brief Title: Pleth Variability Index as a Predictor for Post-induction Hypotension in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Assistant Professor of Anesthesia, SICU & pain management. Kasralainy Faculty of medicine, Cairo University
Other Study IDs: N-126-2020
Record Dates: First submitted 2021-04-13; First posted 2021-05-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Post-induction Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pleth variability index for prediction of post-induction hypotension — The use of the baseline Pleth variability index values for prediction of occurrence of post-induction hypotension

SUMMARY:
Hypotension after induction of general anesthesia and before surgical stimulation is a prevalent anesthesia-related side effect. The post-induction hypotension disrupts organ perfusion and may cause organ damage particularly acute kidney injury, cerebrovascular stroke, and myocardial ischemia. Post-induction hypotension occurs with greater frequency and severity in the elderly. This is because of aged-related diminished cardiac reserve and impaired autonomic homeostasis. Pleth variability index (PVI) is a software program that measures the dynamic changes of the PI that occurs during a complete respiratory cycle. Our primary outcome is to determine the predictive ability and the optimal cut-off value of pre-anesthesia PVI for predicting elderly patients who are at risk of developing post-induction hypotension

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA physical status I or II
* patients will receive general anesthesia

Exclusion Criteria:

* Patients with a history of cardiorespiratory disorders
* patients with uncontrolled hypertension or cardiac dysrhythmias
* Patients with renal or hepatic diseases.
* Patients with long-standing diabetes and peripheral vascular diseases.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: all patients. Patients ≥ 65 years, ASA physical status I or II, and scheduled for elective surgery under general anesthesia will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
The accuracy (Area under receiver operating characteristic curves) of pre-induction PVI for prediction of post-induction hypotension | before induction of general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Abeer Ahmed Mohamed, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided